CLINICAL TRIAL: NCT02392065
Title: Chronic Obstructive Pulmonary Disease as a Predictor of 2-year Mortality in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Chronic Obstructive Pulmonary Disease as a Predictor of Mortality in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: COPD14_2014
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiac Surgery
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To estimate prevalence of chronic obstructive pulmonary disease (COPD) in cardiac surgery population and establish links between COPD status, as assessed through pulmonary functional tests, and 2-year mortality

ELIGIBILITY:
Inclusion Criteria:

* written informed consent, planned elective coronary artery bypass graft surgery

Exclusion Criteria:

* contraindications to pulmonary functional tests, emergency surgery, recent or ongoing myocardial infarction, angina

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for coronary artery bypass surgery during one year will be screened and approached
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lomivorotov, MD, PhD, Study Director — Novosibisrk Research Institute of Circulation Pathology
Locations (1):
- Novosibirsk Research Institute of Circulation Pathology, Novosibirsk, Russia